CLINICAL TRIAL: NCT00571506
Title: A Pilot Study to Determine the Effects of Short-term Thiazolidinedione Treatment on Vascular Risk Markers in Type 2 Diabetes Patients
Brief Title: Effect of Thiazolidinedione Treatment Vascular Risk Markers
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Arkansas (Other)
Responsible Party: Amy M. Franks, Pharm.D., University of Arkansas for Medical Sciences College of Pharmacy
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 26963
Record Dates: First submitted 2007-12-10; First posted 2007-12-12 (Estimated); Last update posted 2009-12-09 (Estimated); Status verified 2009-12

CONDITIONS: Diabetes Mellitus, Type 2; Vascular Diseases
Keywords: Diabetes Mellitus, Type 2; Vascular Diseases; Thiazolidinediones; Platelet Aggregation
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Vascular Diseases | interventions — Rosiglitazone; Pioglitazone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Rosiglitazone 4 mg by mouth daily
  Interventions: Drug: Rosiglitazone
- 2 (Active Comparator): Pioglitazone 30 mg by mouth daily
  Interventions: Drug: Pioglitazone

INTERVENTIONS:
Drug: Rosiglitazone — Rosiglitazone 4 mg tablets by mouth daily for 3 months
  Other Names: Avandia
  Arms: 1
Drug: Pioglitazone — Pioglitazone 30 mg tablet by mouth once daily
  Other Names: Actos
  Arms: 2

SUMMARY:
The purpose of this study is to examine the effects of two diabetes medications, rosiglitazone and pioglitazone, on markers of vascular disease in subjects with type 2 diabetes.

DETAILED DESCRIPTION:
Diabetes is a common disease in the United States, affecting over 10 million Americans. Vascular disease, including heart attack and stroke, affects many diabetic patients and will cause the death of three-fourths of these patients. Because the majority of diabetic patients will suffer complications or death from vascular disease, we will explore treatments that have the potential to reduce or prevent vascular disease in type 2 diabetes patients. Our study will examine the effects of two diabetes medications, rosiglitazone (ROSI) and pioglitazone (PIO), on markers of vascular disease in 20 subjects with type 2 diabetes. It is thought that these two medications will reduce the risk of vascular disease by affecting the platelets and proteins that that regulate the processes involved in clot formation. One-half of the subjects enrolled in our study will take ROSI and the other half will take PIO. We will measure the clumping ability of these subjects' platelets before, during, and after three months of treatment with ROSI or PIO. We will measure the blood concentrations of several proteins (fibrinogen, PAI-1, CRP, adiponectin, and leptin) before and after treatment with the study drugs. These experiments will give us information about any beneficial effects of ROSI and PIO on the clot-forming ability in diabetes patients. We expect that treatment with ROSI and PIO will result in improvement of the disturbed clot-forming processes that predispose diabetic patients to vascular disease.

ELIGIBILITY:
Inclusion Criteria:

* Men and women of all races
* Age 40-65 years
* Diagnosis of type 2 diabetes
* hemoglobin A1C ≥ 7%
* eligible whether or not currently taking antihyperglycemic medications

Exclusion Criteria:

* History of rosiglitazone or pioglitazone use in the previous 3 months
* Known diagnosis of peripheral vascular disease or cardiac failure
* Recent history (within past 6 months) of ischemic stroke, myocardial infarction, percutaneous coronary intervention, or coronary artery bypass surgery
* Active liver disease or elevated serum transaminases (ALT >2.5x upper limit of normal)
* Current therapy with oral anticoagulants (warfarin, heparin, low molecular weight heparin), clopidogrel, or immunosuppressive agents
* Pregnancy or breastfeeding
* Any other condition, in the opinion of the investigator, that renders the subject unable to complete the study, that interferes with optimal participation in the study, or that produces significant risk to the subject

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2004-05; Primary Completion 2007-08 (Actual); Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
determine if treatment with rosiglitazone or pioglitazone affects platelet function as assessed by spontaneous and agonist-induced platelet aggregation | 3 months

SECONDARY OUTCOMES:
adipocytokine concentrations (adiponectin, leptin), hemostatic parameters (fibrinogen, plasminogen activator inhibitor-1), high-sensitivity C-reactive protein | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Amy M. Franks, Pharm.D., Principal Investigator — University of Arkansas
Locations (1):
- University of Arkansas for Medical Sciences, Little Rock, Arkansas, United States